CLINICAL TRIAL: NCT01857661
Title: The Influence of the Sound Generator Combined With Conventional Amplification for Tinnitus Control: Blind Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Gisele Munhoes dos Santos, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/03001-2
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-05

CONDITIONS: Tinnitus; Hearing Loss
Keywords: tinnitus; hearing loss; hearing devices
MeSH Terms: conditions — Tinnitus; Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Other): hearing aid without an integrated sound generator
  Interventions: Device: hearing aids with only amplification
- sound generator (Experimental): hearing aid with an integrated sound generator
  Interventions: Device: sound generator

INTERVENTIONS:
Device: sound generator — hearing aid with an integrated sound generator
  Arms: sound generator
Device: hearing aids with only amplification
  Arms: control

SUMMARY:
The University of Sao Paulo Department of Otorhinolaryngology developed prototypes for a digital new hearing aid with an integrated sound generator. These prototypes assist both hearing rehabilitation (about 10% of the population) and tinnitus sufferers (about 17% of the population).

Currently, the Brazilian Public Heath Care does not have any such hearing aids. So, the development of devices for the hearing rehabilitation as well as the treatment of tinnitus represents an advance in the implementation of Public Policies in Brazil.

The aim of this study is to compare the efficacy of the hearing aid with an integrated sound generator and amplification alone for tinnitus control in patients with tinnitus associated hearing loss.

DETAILED DESCRIPTION:
This study, in the form of a blind randomized clinical trial, was approved by CAPPesq under protocol number: 0163/10.

49 adults with tinnitus and sensorineural hearing loss were randomly assigned into 2 groups. Both groups received counseling about tinnitus. One group received hearing aids with only amplification and the other group received hearing aids with an integrated sound generator. After the fitting process, both groups were told to use the hearing devices 8 hours per day. The outcome measures as the tinnitus handicap inventory and psychoacoustics measurements were conducted by a blind audiologist that didn't know each group each patient belonged to.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate sensorineural hearing loss
* tinnitus (THI > 20)
* first user

Exclusion Criteria:

* profound hearing loss
* conductive hearing loss
* THI < 20

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
THI | 3 months
  tinnitus handicap inventory

REFERENCES:
- [Derived] dos Santos GM, Bento RF, de Medeiros IR, Oiticcica J, da Silva EC, Penteado S. The influence of sound generator associated with conventional amplification for tinnitus control: randomized blind clinical trial. Trends Hear. 2014 Jul 23;18:2331216514542657. doi: 10.1177/2331216514542657. PMID 25073131